CLINICAL TRIAL: NCT00605254
Title: Brain and Whole Body Imaging of P-Glycoprotein Function Using [11C]dLop
Brief Title: PET Imaging of P-glycoprotein Function Using [11C]dLop
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080062; 08-M-0062
Record Dates: First submitted 2008-01-26; First posted 2008-01-31 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-09-04

CONDITIONS: Healthy
Keywords: P-Glycoprotein; Positron Emission Tomography; Blood Brain Barrier; Quantitative Imaging; Multi-Drug Transporter; Healthy Volunteer; HV

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
This study will test the use of a radioactive substance called [11C]dLop for measuring P-glycoprotein (P-gp) using positron emission tomography (PET) imaging. The P-gp protein acts as a pump in cells, affecting a variety of functions, such as limiting drug absorption and elimination and decreasing drug penetration into certain tissues, such as the brain. It is a major obstacle to successful chemotherapy because it can pump cancer drugs out of the cells, interfering with treatment. Decreased P-gp function may contribute to disorders such as Parkinson s disease and Alzheimer s disease, whereas higher levels of the protein have been found in patients with epilepsy and in several forms of drug-resistant cancer tumors. This study will determine uptake and clearance of [11C]dLop and the radiation exposure to organs of the body to assess its possible use in further studies of P-gp function.

Healthy normal volunteers between 18 and 51 years of age may be eligible for this study. Candidates are screened with a medical history, physical examination and blood and urine tests.

Participants undergo the following procedures:

* Electrocardiogram (ECG): A test of the electrical function of the heart.
* Brain PET scans: PET imaging uses small amounts of a radioactive chemical called a tracer that labels active areas of the brain so the activity can be seen with a special camera. The tracer used in this study is [18F]FMPEP-d(2). Before starting the scan, a catheter (plastic tube) is placed in a vein in the arm to inject the tracer and another catheter is placed in an artery in the wrist to obtain blood samples during the scan. For the procedure, the subject lies on the scanner bed. A special mask is fitted to the head and attached to the bed to help keep the person s head still during the scan so the images will be clear. A brief scan is done just before the tracer is injected to provide measures of the brain that are helpful in calculating information from subsequent scans. After the tracer is injected, pictures are taken for about 2.5 hours, while the subject lies still on the scanner bed. Blood and urine tests are done after 24 hours after the scan.
* Magnetic resonance imaging (MRI): An MRI scan is done within 1 year (before or after) of the PET scan. This procedure uses a magnetic field and radio waves to produce images of the brain. The subject lies on a table that is moved into the scanner (a tube-like device), wearing earplugs to muffle the noise of the machine during the scanning process. The test takes about 1 hour....

DETAILED DESCRIPTION:
P-glycoprotein (P-gp) is an ATP-binding cassette (ABC) transporter and is the major efflux pump in the blood-brain barrier. P-gp has several physiological roles such as limiting drug absorption, active drug elimination, and limits drug penetration into sensitive tissues (e.g., brain and testis) (Fromm, 2004). Reduced activity or expression of P-gp may contribute to neurodegenerative disorders such as Parkinson s and Alzheimer s disease. The reduced activity of P-gp (i.e., decreased neuroprotection at the blood brain barrier) may allow harmful pesticides access to the brain which can damage the brain s dopaminergic cell groups possibly leading to Parkinson s disease (Betarbet et al., 2000; Kortekaas et al., 2005). The increased deposition of beta-amyloid in Alzheimer s disease, may be due in part, to the decreased elimination of cerebral beta-amyloid in brain (Vogelgesang et al., 2002). Conversely, an overexpression of P-gp has been found in epilepsy and in several forms of multi drug resistant cancer tumors (Brandt et al., 2006; Szakacs et al., 2006). In vivo evaluation of P-gp function in the brain and throughout the body is important in disease states, and in therapeutic and diagnostic drug evaluation.

P-gp function has been assessed in healthy volunteers with positron emission tomography (PET) using [11C]verapamil, nevertheless, accurate quantification of this PET radioligand is difficult due to the large contribution of radiometabolites and low signal (Ikoma et al., 2006; Lee et al., 2006; Lubberink et al., 2007). Therefore, we have recently developed [11C]dLop as an alternative radioligand for imaging P-gp function, which will allow a more accurate quantification of P-gp with a higher signal and less contribution of radiometabolites. In the current protocol, we wish to evaluate [11C]dLop in healthy volunteers to determine the kinetics of brain imaging of P-gp function. In order to simulate P-gp dysfunction in healthy volunteers we will administer the P-gp inhibitor tariquidar. We will perform brain PET scans using [11C]dLop before and after P-gp blockade in order to quantify P-gp function at the blood-brain barrier.

ELIGIBILITY:
* DESCRIPTION OF STUDY POPULATIONS:

For the dose escalation study using oral tariquidar, we will select healthy adult female and male volunteers (age 18-51 years old). These healthy volunteers will be medication free, excluding birth control pills. These subjects will be asked to abstain from any medications 16 days before and 1 week after participation in the study.

For the AD study, we will select male and female AD patients and age-matched volunteers who are at least 45 years of age.

INCLUSION CRITERIA:

1. Patients with the diagnosis of probable Alzheimer disease. All patients must meet capacity criteria to consent to research (see Consent documents and process).
2. Healthy volunteers.

EXCLUSION CRITERIA:

1. Current psychiatric disease, illicit substance use, or severe systemic disease based on history and physical exam.
2. Laboratory tests with clinically significant abnormalities. Normal organ and marrow function are defined as: total leukocyte count greater than or equal to 3000 cells/ul, ANC greater than or equal to 1500 cells/ul, platelet count greater than or equal to 100,000 cells/ul, serum creatinine less than or equal to 2.0 times the upper limit of normal, and bilirubin less than or equal to 1.5 times the upper limit of normal, hemoglobin 9.0 g/dL , serum calcium less than or equal to 12.0 mg/dL, AST/ALT less than or equal to 1.5 times the upper limit of normal, PT less than or equal to 1.5 times the upper limit of normal.
3. Prior participation in other research protocols or clinical care in the last year such that radiation exposure including that from this protocol would exceed the guidelines set by the Radiation Safety Committee (RSC).
4. Pregnancy or breast feeding.
5. Positive HIV test.
6. Positive result on urine screen for illicit drugs.
7. You cannot lie on your back for extended periods of time.
8. Use of blood-thinning medications (such as warfarin; aspirin is allowed), current or prior history of coagulopathy. This will be necessary only for subjects who have arterial catheter placement.
9. History of neurological disease other than Alzheimer disease.
10. For oral tariquidar dose-escalation study: Subjects taking medications other than birth control pills.
11. For Alzheimer s disease patients and age-matched volunteers: Subjects taking medications that are known substrates of P-gp that cannot be safely discontinued for this study.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2008-01-24; Study Completion 2014-09-04

PRIMARY OUTCOMES:
PET | continuous

CONTACTS AND LOCATIONS:
Overall Officials: William C Kreisl, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Awouters F, Niemegeers CJ, Janssen PA. Pharmacology of antidiarrheal drugs. Annu Rev Pharmacol Toxicol. 1983;23:279-301. doi: 10.1146/annurev.pa.23.040183.001431. No abstract available. PMID 6307123
- [Background] Betarbet R, Sherer TB, MacKenzie G, Garcia-Osuna M, Panov AV, Greenamyre JT. Chronic systemic pesticide exposure reproduces features of Parkinson's disease. Nat Neurosci. 2000 Dec;3(12):1301-6. doi: 10.1038/81834. PMID 11100151
- [Background] Bigott HM, Prior JL, Piwnica-Worms DR, Welch MJ. Imaging multidrug resistance P-glycoprotein transport function using microPET with technetium-94m-sestamibi. Mol Imaging. 2005 Jan-Mar;4(1):30-9. doi: 10.1162/15353500200504166. PMID 15967124
- [Derived] Kreisl WC, Bhatia R, Morse CL, Woock AE, Zoghbi SS, Shetty HU, Pike VW, Innis RB. Increased permeability-glycoprotein inhibition at the human blood-brain barrier can be safely achieved by performing PET during peak plasma concentrations of tariquidar. J Nucl Med. 2015 Jan;56(1):82-7. doi: 10.2967/jnumed.114.146894. Epub 2014 Dec 11. PMID 25500831